CLINICAL TRIAL: NCT04596397
Title: Oral Misoprostol for Outpatient Induction of Labor; a Pilot Randomized-controlled Trial
Brief Title: Oral Misoprostol for Outpatient Induction of Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020/104044
Record Dates: First submitted 2020-10-12; First posted 2020-10-22 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Labor Induction
Keywords: induction of labor; outpatient setting; misoprostol

STUDY DESIGN:
Intervention Model Description: All eligible women will be recruited form a midwife and/or doctor. After the inclusion they will be randomized to either inpatient or outpatient setting.
Masking Description: The women included will be randomized from number 1 -20 where number 1-10 are inpatient and number 11-20 are outpatient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Induction of labour with oral misoprostol, inpatient setting (Active Comparator): These women receive all treatment in the maternity unit.
  Interventions: Other: Inpatient setting
- Induction of labour with oral misoprostol, outpatient setting (Experimental): These women will be observed 2 hours after they receive one dose of oral misoprostol before the can leave the maternity unit.
  Interventions: Other: Outpatient setting

INTERVENTIONS:
Other: Inpatient setting — These women stay at the hospital.
  Arms: Induction of labour with oral misoprostol, inpatient setting
Other: Outpatient setting — These women can leave the hospital.
  Arms: Induction of labour with oral misoprostol, outpatient setting

SUMMARY:
An increasing proportion of pregnant women have their labors induced due to changing guidelines. In correlation with this increase, the population of the induced women has changed toward more women with a low-risk pregnancy. Traditionally, induction of labor has taken place in an inpatient setting where the women have spent extra days in hospital before delivery.

Oral prostaglandins, such as misoprostol, is one of the most commonly used induction agent and is easy for the pregnant women to administrate. The pharmacological effect is ripening the cervix and compared to the mechanical cervical ripening, with a balloon catheter, the demands on busy maternity services seems reduced. Before contractions start, the risk of adverse effects on mother or fetus is considered low, but the evidence on use of misoprostol in an outpatient setting is sparse.

DETAILED DESCRIPTION:
The implementation of induction of labor in outpatient settings is increasing despite insufficient evidence regarding safety and effectiveness. The use of a balloon catheter in an outpatient setting is not associated with adverse outcomes in a low-risk population. There is also evidence that outpatient vs inpatient induction of labor with balloon catheter is equally effective. Examination of vaginal dinoprostone (prostaglandin E2) is found to be efficacious in outpatient settings. However, strong evidence concludes that the oral route of administration of prostaglandin is preferable when inducing labor. The World Health Organization recommend 25ug misoprostol (prostaglandin E1) orally every 2 hour until contractions start for induction of labor.

The women randomized to an inpatient setting will receive the hospital standard follow-up; oral misoprostol 25ug every two hours and a cardiotocography for fetal monitoring every 4-6 hour until start of contractions for two days.

The women randomized to an outpatient setting will receive one oral misoprostol 25ug at the maternity unit. After two hours, provided a normal cardiotocography and no contractions, they can go home. They will continue to take 25ug misoprostol every two hours until start of contractions or increasing pain. Maximum time spent at home will be 48 hours.

A dedicated midwife on call will always be available for questions. The women will receive oral and written information to return to the maternity unit if the water breaks, if they experience increasing pain or bleeding, if they feel insecure or anxious, if there are reduced or no fetal movements, and/or when the contraction starts. When the woman returns, she will stay admitted until delivery.

All women will be given standard of care and fetal surveillance when admitted to the hospital, when the contractions start or if the contractions are still absent after 48 hours. We will also ask eligible women who refrain to participate about their reasons for non-participation.

PRIMARY RESEARCH QUESTION We aim to explore that induction of labor using oral misoprostol appears feasible in an outpatient setting and may positively influence the length of the hospital stay and maternal satisfaction.

PRIMARY RESEARCH PLAN This is a pilot study to explore the feasibility of a possible multicenter randomized controlled trail.

ELIGIBILITY:
Inclusion Criteria:

* Understand and read Norwegian
* No cognitive barriers. The woman must be able to give informed consent
* ≥ 37 gestational week, vertex presentation, single pregnancy
* Normal ultrasound including fetal movements, amniotic fluid, estimated fetal weight +/- 15% (≤ 10 percentile and ≥ 90) and normal doppler peak systolic index in the umbilical cord artery and the cerebri media artery
* Normal cardiotocography
* Body Mass Index 18-35
* No signs of infection or health problems
* Distance to hospital 45-60 minutes

Exclusion Criteria:

* Premature rupture of membranes
* Previous cesarean section or operation on uterus
* Fetal anomaly or chromosome/genetic disorder
* Pregnancy complications such as preeclampsia and diabetes (insulin dependent) or other conditions were changes in fetal heart rate during labor is suspected
* Not eligible for misoprostol as induction agent due a favorable cervix (Bishop score) and/or previous obstetric history

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
The feasibility of a randomised controlled trial of outpatient labor induction | 6 months
  The number of eligible women who is willing to enrol in participating

SECONDARY OUTCOMES:
Reported labor experience among the women participating | From included in the study until postpartum discharge (1-2 weeks)
  The women will fill out a survey before and after birth (including childbirth expectations, experience and satisfaction)
Maternal length of hospital stay | From included in the study until postpartum discharge (1-2 weeks)
  Length of hospital stay form start of induction to postpartum discharge
Use of analgesia | From start of the partogram until birth (hours)
  Use of epidural and fentanyl analgesia during labor

CONTACTS AND LOCATIONS:
Overall Officials: Janne Rossen, MD, PhD, Principal Investigator — Sorlandet Hospital Trust, Kristiansand, Norway
Locations (1):
- Sorlandet Hospital Trust, Kristiansand, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vogel JP, Osoti AO, Kelly AJ, Livio S, Norman JE, Alfirevic Z. Pharmacological and mechanical interventions for labour induction in outpatient settings. Cochrane Database Syst Rev. 2017 Sep 13;9(9):CD007701. doi: 10.1002/14651858.CD007701.pub3. PMID 28901007
- [Background] Alfirevic Z, Aflaifel N, Weeks A. Oral misoprostol for induction of labour. Cochrane Database Syst Rev. 2014 Jun 13;2014(6):CD001338. doi: 10.1002/14651858.CD001338.pub3. PMID 24924489
- [Background] WHO Recommendations for Induction of Labour. Geneva: World Health Organization; 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK131963/ PMID 23586118
- [Background] Diederen M, Gommers J, Wilkinson C, Turnbull D, Mol B. Safety of the balloon catheter for cervical ripening in outpatient care: complications during the period from insertion to expulsion of a balloon catheter in the process of labour induction: a systematic review. BJOG. 2018 Aug;125(9):1086-1095. doi: 10.1111/1471-0528.15047. Epub 2018 Jan 10. PMID 29211328
- [Background] Wilkinson C, Bryce R, Adelson P, Turnbull D. A randomised controlled trial of outpatient compared with inpatient cervical ripening with prostaglandin E(2) (OPRA study). BJOG. 2015 Jan;122(1):94-104. doi: 10.1111/1471-0528.12846. Epub 2014 May 14. PMID 24824157